CLINICAL TRIAL: NCT03322501
Title: Pediatric Health Promotion Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-0787
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The purpose of the study is to determine if an Ask, Advise, Connect (AAC) intervention model benefits tobacco control outcomes for pediatric primary care providers (pPCP's) and their young patients.
  Interventions: Behavioral: Provider Advice, Framed Messaging

INTERVENTIONS:
Behavioral: Provider Advice, Framed Messaging — The purpose of the study is to determine if an Ask, Advise, Connect (AAC) intervention model benefits tobacco control outcomes for pediatric primary care providers (pPCP's) and their young patients.

SUMMARY:
The purpose of the study is to determine if an Ask, Advise, Connect (AAC) intervention model benefits tobacco control outcomes for pediatric primary care providers (pPCP's) and their young patients.

ELIGIBILITY:
Inclusion Criteria:

* Well-child visit

Exclusion Criteria:

-

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Tobacco Use | 1 Month

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No